CLINICAL TRIAL: NCT03883997
Title: Accuracy of Anthropometric Equations for Estimating Body Fat in Professional Male Soccer Players Compared With DXA
Status: Completed | Type: Observational
Sponsor: Centro Universitario de Ciencias de la Salud, Mexico (Other)
Responsible Party: Principal Investigator, Juan Ricardo Lopez y Taylor, Director of the Institute of Applied Sciences for Physical Activity and Sport, Centro Universitario de Ciencias de la Salud, Mexico
Other Study IDs: LNFUT-1
Record Dates: First submitted 2019-03-19; First posted 2019-03-21 (Actual); Last update posted 2019-03-21 (Actual); Status verified 2019-03

CONDITIONS: Body Composition
Keywords: Body fat; Soccer players; DXA

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Participants: Professional male soccer players from the second professional Mexican division.
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — Cross-sectional

SUMMARY:
This study aimed to analyze the accuracy of different anthropometric equations to estimate body fat in professional male soccer players, setting DXA body fat as the reference.

DETAILED DESCRIPTION:
The study consisted of evaluating anthropometric measurements and body composition with DXA in professional male soccer player aged 18 years and older. Standardized and certified personnel carried out anthropometric measurements and DXA whole body scan the same day.

Body fat was estimated with several anthropometric equations. These equations were divided into two groups: 1) Derived from non-athletic samples; and 2) Derived from athletic samples.

The body fat estimated from anthropometric equations was compared with DXA, and those with non-significant differences were further analyzed for calculating mean differences and 95% limits of agreement with DXA. This analysis was carried out for all equations.

ELIGIBILITY:
Inclusion Criteria:

* Signed contract with the team

Exclusion Criteria:

* Injured

Ages: 18 Years to 37 Years | Sex: Male
Age Groups: Adult
Study Population: Professional male soccer players hired into a second professional Mexican division team.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2009-08 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2018-01 (Actual)

PRIMARY OUTCOMES:
Body fat by DXA | One day
  Body fat obtained from a whole body DXA scan transformed from grams to percentage.

CONTACTS AND LOCATIONS:
Overall Officials: Juan R López-Taylor, Study Director — University of Guadalajara
Locations (1):
- Instituto de Ciencias Aplicadas a la Actividad Física y al Deporte, Guadalajara, Jalisco, Mexico

IPD SHARING:
Plan to Share IPD: Undecided